

# T.C ESKİŞEHİR OSMANGAZİ ÜNİVERSİTESİ KLİNİK ARAŞTIRMALAR ETİK KURULU (LOCAL ETHIC BOARD-STUDY PROTOCOL)

Version date: 15/07/2017 Version number: 1

TITLE: Superior Rectal Artery Embolization With Tri-acryl Gelatin Particles for Treatment of Symptomatic Hemorrhoids: Safety and Efficacy

## Principle investigator-coordinator (\*\*):

Prof.Dr.Fahrettin Küçükay (\*\*)

# **Investigators:**

Assoc.Prof.Dr. Necdet Fatih Yaşar

Ass.Prof.Dr.Bartu Badak

Assoc.Prof. Dr. Tuncer Temel

Location: Eskisehir Osmangazi University, Faculty of Medicine, Interventional Radiology,

Gastroenterology, General Surgery, Eskisehir/Turkey

**Study design:** Double arm, parallel, single blinded, blocked randomized ,prospective study

**Unique Protocol ID:** 80558721/237

#### INTRODUCTION

Symptomatic hemorrhoidal disease is a still important public health problem although there are many surgical and nonsurgical minimal invasive treatment methods. Treatment methods are not satisfactory or invasive in some percent of the patients. Superior rectal artery embolization (SRAE) for hemorrhoids is an adapted technique derived from Doppler-guided hemorrhoidal artery ligation (DGHAL). In this technique, the distal branches of the superior rectal artery arising from the inferior mesenteric artery is occluded endovascularly with coils. Its feasibility and safety were supported by articles. Collateralization and recurrence was seen following coil embolization.

<sup>13</sup> Nisan 2013 tarih ve 28617 sayılı Resmi Gazetede yayınlanan İlaç Ve Biyolojik Ürünlerin Klinik Araştırmaları Hakkında Yönetmelik:

<sup>(\*)</sup> y) Sorumlu araştırmacı: Araştırma konusu ile ilgili dalda uzmanlık veya doktora eğitimini tamamlamış olup, araştırmanın yürütülmesinden sorumlu olan hekim veya diş hekimini,

<sup>(\*\*)</sup> cc) (Ek:RG-25/6/2014-29041) <u>Koordinatör:</u> Çok merkezli bir araştırmada bu merkezlerin sorumlu araştırmacıları ile etik kurul, destekleyici veya destekleyicinin yasal temsilcisi ve gerekirse bunlar ile Kurum arasındaki koordinasyonun sağlanmasından sorumlu, uzmanlığını veya doktorasını tamamlamış hekim veya diş hekimini,

The purpose of this study is to compare safety and efficacy of 500-700 and 700-900 micron microspheric particles in superior rectal artery embolization.

## **MATERIALS AND METHODS**

This is a double arm, parallel, single blinded, blocked randomized, prospective study. In each arm there will be 25 patients (any sex, between 18-75 years old). Local ethic board approved the study. Written informed consent will be obtained from the patients included in the study. Study will be conducted between December 2018 and Deecember 2019.

Inclusion criteria as follows:

- -Patients with symptoms of hemorrhoidal disease
- Patients with written informed consent
- Patients refusing surgery or other interventional methods
- Patients with high risk for surgery
- Patients accepting follow ups

Exclusion criteria as follows:

- Previous intervention
- Colorectal diseases other than hemorrhoids
- -Patients with anal stenosis
- Patients with rectal prolapsus
- pregnant patients
- Patients with contraindications for technical steps or contrast usage.
- -Patients do nor or could not give written informed consent

In experimental arms interventional embolization with 500-700 and 700-900 micron particles will be performed with 1 ml vials. Embolization procedure will be continued with vials until the stasis in SRAE will be achieved. Procedure will be performed only one time.

Primary Outcome Measures are as follow:

- -Incidence of procedure related mortality (safety) [Time Frame: 12 month]. The mortality rate among the patients during 12 months related with interventional procedure.
- Incidence of procedure related complications (safety) [Time Frame: 12 month]. The morbidity rate among the patients during 12 months related with interventional procedure.
- Incidence of the patients' being free of symptoms from hemorrhoidal disease (efficacy) [Time Frame: 12 month]. The efficacy and clinical success of the procedure will be evaluated.

[Metni yazın]

Secondary Outcome Measures:

- -Technical success [Time Frame: On the day of intervention]. The rate of interventions that were performed successfully.
- Recurrence [Time Frame: 3-6-12. months]. Recanalization or collateralization of the previously embolized rectal arteries.

Goligher's classification scale (prolapse stage), Bleeding severity score (French), Qulity of life score, Visual analog scale score for pain will be used for follow ups.

Appropriate statistical analysis of primary and secondary outcomes will be used to describe the results of data obtained.

#### **REFERENCES:**

- 1: Zakharchenko A, Kaitoukov Y, Vinnik Y, Tradi F, Sapoval M, Sielezneff I,Galkin E, Vidal V. Safety and efficacy of superior rectal artery embolization with particles and metallic coils for the treatment of hemorrhoids (Emborrhoid technique). Diagn Interv Imaging. 2016 Nov;97(11):1079-1084. doi: 10.1016/j.diii.2016.08.002. Epub 2016 Aug 31. PubMed PMID: 27597728.
- 2: Vidal V, Sapoval M, Sielezneff Y, De Parades V, Tradi F, Louis G, Bartoli JM, Pellerin O. Emborrhoid: a new concept for the treatment of hemorrhoids with arterial embolization: the first 14 cases. Cardiovasc Intervent Radiol. 2015 Feb;38(1):72-8. doi: 10.1007/s00270-014-1017-8. Epub 2014 Nov 4. PubMed PMID: 25366092.
- 3: Vidal V, Louis G, Bartoli JM, Sielezneff I. Embolization of the hemorrhoidal arteries (the emborrhoid technique): a new concept and challenge for interventional radiology. Diagn Interv Imaging. 2014 Mar;95(3):307-15. doi: 0.1016/j.diii.2014.01.016. Epub 2014 Feb 28. PubMed PMID: 24589187.
- 4: Galkin E. [X-ray endovascular embolization of the superior rectal artery: New potentialities in the surgical management of chronic hemorrhoids]. Vestn Rentgenol Radiol. 2001 Nov-Dec;(6):44-9. Russian. PubMed PMID: 11858033.
- 5: Galkin EV, Iavisia AM, Vdovenko PA. [Interventional radiology for chronic hemorrhoids complicated by hemorrhage]. Vestn Rentgenol Radiol. 1998 Sep-Oct;(5):21-4. Russian. PubMed PMID: 9987939.
- 6: Galkin EV. [Interventional radiology of chronic hemorrhoids]. Vestn Rentgenol Radiol. 1994 Jul-Aug;(4):52-6. Russian. PubMed PMID: 7785199.

### **FLOW-CHART**



PROFESSOR DR FAHRETTIN KÜÇÜKAY,(IR)
ASSISTANT PROFESSOR DR. BARTU BADAK, (GS)
ASSOCIATE PROFESSOR DR. NECDET FATIH YAŞAR,(GS)
ASSOCIATE PROFESSOR DR. TUNCER TEMEL(GE)